CLINICAL TRIAL: NCT06203652
Title: The Pathogenesis and Prognostic Factors of Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Peng Liu, Chief of Hematology department, Shanghai Zhongshan Hospital
Other Study IDs: SHZS-lym-001
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma; Hodgkin Lymphoma; Non-hodgkin Lymphoma
Keywords: lymphoma; Hodgkin lymphoma; Non-Hodgkin lymphoma; THRLBCL; DLBCL; MZL; CLL/SLL; MCL; WM
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All enrolled patients: All patients who are eligible for participation to the study.
  Interventions: Other: Real-world regimen

INTERVENTIONS:
Other: Real-world regimen — The final personalized management strategy is determined based on current conventional treatment options, physician and patient preferences.The following protocols: chemotherapy, immunochemotherapy,Anti-cd20 monoclonal antibody, BTKi and so on

SUMMARY:
The aim of this study is to describe the clinical and genetic characteristics of Chinese lymphoma patients, and to explore the relationship between those characteristics and phatogenesis.

DETAILED DESCRIPTION:
Lymphoma is a highly common malignant tumor in Asia. This study aims to observe and describe the clinical and genetic charateristics of Chinese lymphoma patients, and to explore the relationship between those charateristics and pathogenesis and prognostic factors in the real-world population. This study is a non-interventional real world, observational study and all registered data are collected from real clinical practice cases. The medical data includes patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, efficacy results and possible prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosis of lymphoma (including Hodgkin lymphoma and non-Hodgkin lyphoma, eg. THRLBCL, DLBCL, MZL, CLL/SLL...) from 2007 to 2027.
* Patients with complete diagnostic, treatment and follow-up records.
* Fully comprehension and signature of the informed consent form (ICF) for participation.

Exclusion Criteria:

* Those who refuse to use reliable methods of contraception during pregnancy, lactation or age-appropriate period.
* Severe mental illness.
* Patients deemed unsuitable for inclusion by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathological diagnosis of lymphoma from 2007 to 2027 according to 2016 WHO classification.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | Baseline up to data cut-off (Up to approximately 20 years)
  Overall survival (OS) refers to the time from receiving the first dose to death from any cause

SECONDARY OUTCOMES:
PFS | Baseline up to data cut-off (Up to approximately 20 years)
  Progression-free survival (PFS) is defined as the time from the date of first administration to the date of first disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality, China